CLINICAL TRIAL: NCT03115684
Title: Antalgie à l'Accueil Des Urgences- étude de prévalence
Brief Title: Pain Relief in the Emergency Department Waiting Room: a Prevalence Study
Status: Completed | Type: Observational
Sponsor: University Hospital, Geneva (Other)
Responsible Party: Principal Investigator, Majd Ramlawi, Médecin adjoint du chef de service, University Hospital, Geneva
Other Study IDs: 215-00083-(15-272)
Record Dates: First submitted 2017-04-11; First posted 2017-04-14 (Actual); Last update posted 2017-04-14 (Actual); Status verified 2017-04

CONDITIONS: Acute Pain
MeSH Terms: conditions — Acute Pain

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Pain in the emergency room is under documented and pain relief suboptimal. Data on nurse driven analgesia in emergency department waiting rooms is lacking. The primary objective of this study is to determine the proportion of patients in pain receiving pain therapy administered by the triage nurse (prevalence study). The secondary objectives are to 1) describe nursing practices in analgesia and adherence to the dedicated protocol; 2) to determine the factors associated with the non administration of painkillers and for these factors, to estimate the strength of the association

ELIGIBILITY:
Inclusion Criteria:

* Documented pain score on arrival by the triage nurse and
* Patients having to wait in the ER waiting room

Exclusion Criteria:

* patients directly admitted to the consultation room
* patients for whom pain was not recorded

Min Age: 16 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Patients admited to an emergency department waiting room after triage with a documented pain score upon arrival
Sampling Method: Non-Probability Sample
Enrollment: 2371 (Actual)
Dates: Start 2016-03-01 (Actual); Primary Completion 2016-05-30 (Actual); Study Completion 2016-05-30 (Actual)

PRIMARY OUTCOMES:
Proportion of patients receiving pain medicine in the ER waiting room by the triage nurse after pain documentation | 3 month